CLINICAL TRIAL: NCT07039500
Title: Impact of Severe Obstructive Sleep Apnea-Hypopnea Syndrome on Auditory-Cognitive Processing
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUFH-2024RES651-001
Record Dates: First submitted 2025-06-06; First posted 2025-06-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea; Auditory Processing Disorder
Keywords: Obstructive Sleep Apnea; Auditory Cognition; Electroencephalography (EEG); Oddball Paradigm
MeSH Terms: conditions — Sleep Apnea, Obstructive; Auditory Perceptual Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe OSAHS Group: Adults aged 20-60 years with severe obstructive sleep apnea-hypopnea syndrome (AHI>30 events/hour) confirmed by polysomnography (PSG). Participants undergo PSG, hearing tests (pure-tone audiometry, tympanometry), Montreal Cognitive Assessment (MoCA), and EEG recording during active/passive auditory oddball tasks measuring MMN, P300, and behavioral responses.
- Healthy Control Group: Age/sex-matched healthy adults (20-60 years) with self-reported absence of snoring/sleep disorders. Participants complete hearing tests (pure-tone audiometry, tympanometry), Montreal Cognitive Assessment (MoCA), and EEG recording during identical auditory oddball tasks as the OSAHS group.

SUMMARY:
The goal of this observational study is to learn how severe obstructive sleep apnea-hypopnea syndrome (OSAHS) affects the brain's ability to process sounds and attention in adults aged 20-60 years. The main questions it aims to answer are:

1. Does severe OSAHS change how the brain automatically detects sound changes during wakefulness?
2. Does severe OSAHS reduce people's ability to pay attention to important sounds when awake?
3. Can brainwave tests (Electroencephalogram, EEG) detect early signs of hearing-related cognitive problems in OSAHS patients before symptoms appear?

Researchers will compare two groups:

* 50 adults with severe OSAHS (diagnosed by sleep tests)
* 50 healthy adults matched by age and gender

Participants will:

* Complete hearing tests (MoCA)
* Undergo a 1-night sleep test (PSG)
* Wear an EEG cap for 1.5-2 hours while listening to sounds in a quiet room:

  * Passive task: Relax (no response needed)
  * Active task: Press a button when hearing rare sounds
* Receive ¥75/hour compensation for their time

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Aged 20-60 years
* Normal hearing (PTA ≤25 dB HL at 0.5,1,2,4 kHz; Type A tympanogram)
* MoCA score ≥26
* Willing to complete EEG testing

OSAHS Group Additional:

- PSG-confirmed severe OSAHS (AHI >30 events/hour)

Control Group Additional:

* Self-reported absence of snoring/sleep disorders
* No prior OSAHS diagnosis

Exclusion Criteria:

All Participants:

* History of:

  * Schizophrenia, epilepsy, Parkinson's, TBI, or language disorders
  * Middle/inner ear diseases (otitis media, acoustic neuroma, etc.)
  * Cognitive impairment or depression/anxiety disorders
* Chronic steroid use
* Systemic inflammatory diseases or malignancies
* Pregnancy or suspected pregnancy (self-reported)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two distinct populations:
  1. Severe OSAHS Patients:
     * Recruited from otolaryngology clinics at Peking University First Hospital
     * Diagnosed via in-lab PSG (AHI>30)
  2. Healthy Controls:
     * Community volunteers from Beijing area
     * Age/sex-matched to OSAHS group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Mismatch Negativity (MMN) | Day 1
  EEG-derived MMN amplitude (microvolts, μV) during oddball task. Lower values indicate impaired automatic sound change detection.
Latency of Mismatch Negativity (MMN) | Day 1
  EEG-derived MMN latency (milliseconds, ms) during oddball task. Longer values indicate slower automatic processing.

SECONDARY OUTCOMES:
Reaction Time in Active Auditory Oddball Task | Day 1
  Time taken to press button after deviant sound onset (milliseconds). Higher values indicate slower processing speed.
Accuracy in Active Auditory Oddball Task | Day 1
  Percentage of correct button presses to deviant sounds (%). Lower values indicate worse performance.
Inter-Trial Phase Coherence (ITPC) in Theta/Alpha/Beta Bands | Day 1
  EEG oscillatory synchronization (range 0-1; 0=no phase consistency). Lower values indicate neural desynchronization during auditory processing.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China